CLINICAL TRIAL: NCT03205111
Title: Endometrial Characterization Using Office Hysteroscopy in Women Presenting With Abnormal Uterine Bleeding
Brief Title: Role of Office Hysteroscope in Premenopausal Uterine Bleeding
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Zaki Fahmi, Dr, Assiut University
Other Study IDs: Office Hysteroscope
Record Dates: First submitted 2017-06-29; First posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Uterine Bleeding
MeSH Terms: conditions — Uterine Hemorrhage

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to photographically characterize the endometrium in patients presenting with abnormal uterine bleeding at age group from 20 to 45 years old.

and compare dilatation and curettage with hysteroscopy in obtaining an accurate diagnosis of the etiology of abnormal uterine bleeding.

DETAILED DESCRIPTION:
Menstrual dysfunction is the cause of discomfort and disturbed healthy lifestyle. Abnormal uterine bleeding (AUB) is considered as a common problem in premenopausal women. AUB is defined as bleeding from the uterine that is abnormal in volume, regularity, and/or timing.

There are various diagnostic modalities available in the market, ranging from traditional dilation and curettage (D&C), transvaginal sonography, hysteroscopy and saline infusion sonography. Dilation and curettage is the most widely used simple day care procedure for histological evaluation of the endometrial. It was once considered as the gold standard of investigating women with AUB.

Office hysteroscopy is a very useful technique for diagnosis and treatment of uterine pathology in an office-based environment. It is directly related to the technological explosion, which during the last years has further evolved and given us the opportunity to perform hysteroscopy without providing general anesthesia or sedation to the patients, due to the narrow width of the latest generation hysteroscopes. Hysteroscopic inspection of uterine cavity is a simple and well accepted method. The direct real time visualization, real-color, hydrated, well-illuminated, and augmented vision of the uterine cavity make this diagnostic tool very accurate to detect minute focal endometrial pathology and small lesions and helping us to take well guided direct biopsies.

ELIGIBILITY:
Inclusion Criteria:

* Perimenopausal women complaining of abnormal uterine bleeding.

Exclusion Criteria:

* Active pelvic infections
* Medical disorders
* Bleeding tendency
* Hormonal treatment
* Pregnancy
* Contraceptive treatment

Ages: 20 Years to 45 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: 100 women between 20 and 45 years of age who presented with complaints of abnormal uterine bleeding will be recruited for this study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-07 (Estimated); Primary Completion 2018-06 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Hysteroscopic assessment of endometrial pathology | 7 days
  Patterns of endometrial pathology after histopathological examination of the curretings in patients with abnormal uterine bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Z. Fahmi, Principal Investigator — Assiut University; Essam M. Abdallah, Profosser, Study Chair — Assiut University; Hazem S. Mohammed, Professor, Study Director — Assiut University; Kamal M. Zahran, Professor, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bennett AR, Gray SH. What to do when she's bleeding through: the recognition, evaluation, and management of abnormal uterine bleeding in adolescents. Curr Opin Pediatr. 2014 Aug;26(4):413-9. doi: 10.1097/MOP.0000000000000121. PMID 25007322
- [Result] Saadia A, Mubarik A, Zubair A, Jamal S, Zafar A. Diagnostic accuracy of endometrial curettage in endometrial pathology. J Ayub Med Coll Abbottabad. 2011 Jan-Mar;23(1):129-31. PMID 22830167
- [Result] Zhu HL, Liang XD, Wang JL, Cui H, Wei LH. Hysteroscopy and directed biopsy in the diagnosis of endometrial carcinoma. Chin Med J (Engl). 2010 Dec;123(24):3524-8. PMID 22166624